CLINICAL TRIAL: NCT04614987
Title: Serum Neurofilament Light (NfL) as a Marker for Brain Injury in Individuals Undergoing Chimeric Antigen Receptor-modified T Therapy
Status: Terminated | Type: Observational
Why Stopped: PI decided to close study early.
Sponsor: Washington University School of Medicine (Other)
Collaborators: McDonnell Center (Unknown); Paula and Roger Riney Blood Cancer Research (Unknown); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 202009118; K12CA167540 (NIH)
Record Dates: First submitted 2020-10-07; First posted 2020-11-04 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Neurotoxicity
MeSH Terms: conditions — Neurotoxicity Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants undergoing CAR T transfusion: Participants will undergo baseline examination followed by evaluations between Days 3 and 5 post-transfusion, on Day 30 post-transfusion date (PTD), PTD 90, and PTD 180. At baseline this will include plasma testing, lumbar puncture (voluntary), neuroimaging (voluntary) and neuropsychiatric performance testing (voluntary). Between post-transfusion Day 3 and day 5, participants will undergo repeat exam, plasma testing, lumbar puncture (voluntary), and neuroimaging (voluntary). Day 30 testing will again test all modalities, including serum, CSF/lumbar puncture (voluntary), brain imaging (voluntary), and formal neuropsychiatric performance testing (voluntary). Finally, Day 90 and 180 will repeat serum testing, brain imaging, and formal neuropsychological performance testing.

SUMMARY:
The investigators propose that immune effector cell-associated neurotoxicity syndrome (ICANS) is predicated upon the early loss of blood brain barrier (BBB) integrity with subsequent monocyte infiltration leading to cross-activation of native glial cells. Glial overstimulation leads to neuroinflammation, synaptic dysfunction, and ultimately neuronal injury.

ELIGIBILITY:
Inclusion Criteria:

* Clinically scheduled to undergo treatment with tisagenlecleucel, axicabtagene ciloleucel, brexucabtagene autoleucel, or lisocabtagene maraleucel.
* At least 18 years of age.
* Able and willing to undergo study testing (blood draws, lumbar punctures, neuro-psychiatric testing, and neuroimaging with MRI)
* Participants of childbearing potential without documented history of menopause or hysterectomy who choose to participate must not be pregnant at screening and must agree to avoid becoming pregnant prior to scanning.
* Able to understand and willing to sign an IRB-approved written informed consent document.

Exclusion Criteria:

* Has any condition that, in the Investigator's opinion, could increase risk to the participant, limit the participant's ability to tolerate the experimental procedures, or interfere with the collection/analysis of the data (for example, participants unable to lie flat for the duration of the MRI scan).
* Contraindications to MR imaging (e.g. electronic medical devices, inability to lie still for long periods) that make it unsafe for the individual to participate. Patients with pacemakers may only be scanned if approved by CCIR staff and radiology review.
* Severe claustrophobia.
* History of multiple sclerosis, Parkinson's disease, dementia (including Alzheimer's disease, frontotemporal dementia, and Pick's disease), or motor neuron disease including amyotrophic lateral sclerosis (ALS)
* For the lumbar puncture associated with the study only: contraindications to lumbar puncture (e.g. platelets <r 50,000/mm3, INR > 1.5, evidence of midline shift on imaging, presence of local infection at LP site, history of baclofen pump, history of significant spinal surgery/hardware which would preclude safe bedside lumbar puncture). If a contraindication to lumbar puncture develops while on study, patient may remain on study but will be barred from a lumbar puncture until that contraindication resolves.
* Pregnant
* Enrolled in an interventional study of a drug targeting neurotoxicity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants scheduled to undergo treatment at Siteman Cancer Center at Washington University School of Medicine with tisagenlecleucel, axicabtagene ciloleucel, brexucabtagene autoleucel, or lisocabtagene maraleucel.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2021-02-25 (Actual); Primary Completion 2023-09-13 (Actual); Study Completion 2023-09-13 (Actual)

PRIMARY OUTCOMES:
Percent changes in given biomarker levels | From baseline to up to 180 days post-transfusion (estimated to be 7 months)
  * This includes serum (GFAP and NfL) and CSF biomarkers (NfL, VILIP-1, YKL-40, TREM2, and Neurogranin) measured using a single molecule array in pg/ml
  * Descriptive statistics will be used to summarize a given biomarker level at different time points.

SECONDARY OUTCOMES:
Cross-sectional biomarker profiles | From baseline to up to 180 days post-transfusion (estimated to be 7 months)
  -Serum (GFAP, NfL) and CSF biomarkers (NfL, VILIP-1, YKL-40, TREM2, and Neurogranin) as measured using a single molecule array in pg/ml will be compared between participants who develop ICANS compared to participants who do not develop ICANS using descriptive statistics
Cross-sectional imaging profile | From baseline to up to 180 days post-transfusion (estimated to be 7 months)
  -Diffusion basis spectrum imaging (DBSI) separates the point diffusion properties of water by magnitude and direction to provide a non-invasive measurement of cellularity, extracellular edema, and axonal integrity/myelination in μm^2/msec. All three components will then be compared between participants who develop ICANS compared to participants who do not develop ICANS using descriptive statistics
Cytokine profiles | From baseline to up to 180 days post-transfusion (estimated to be 7 months)
  -Elisa-based assays will measure the CSF cytokine profile measurements of IL-2, IL-6, IL10, IFN-y, TNFα, GM-CSF (ng/ml), with descriptive statistics used to compare between participants who develop ICANS compared to participants who do not develop ICANS
Changes in cognitive assessment as measured by Symbol Digit Modalities Test (SDMT) | Baseline, 30 days, 90 days, and 180 days post-transfusion (estimated to be 7 months)
  -The SDMT is a brief written test where participants use a key to match abstract symbols paired with numbers. The scale ranges from 0 to 110, with higher scores reflecting better function. By doing so, an indirect measure of attention, processing speed, motor speed, and visual scanning is obtained. Scores on formal testing will be then be analyzed in conjunction with quantification of imaging features (as parceled using DBSI) observed between participants who develop ICANS compared to participants who do not develop ICANs
Changes in cognitive assessment as measured by Trail Making Test A/B | Baseline, 30 days, 90 days, and 180 days post-transfusion (estimated to be 7 months)
  This brief written test has participants connect lines between sequential numbers and/or letters in a given pattern. By doing so, an indirect measure of executive function tests task switching, visual search, scanning, processing speed, and visual attention is obtained. Scores on formal testing will be then be analyzed in conjunction with quantification of imaging features (as parceled using DBSI) observed between participants who develop ICANS compared to participants who do not develop ICANs
Changes in cognitive assessment as measured by Letter-Number Sequencing | Baseline, 30 days, 90 days, and 180 days post-transfusion (estimated to be 7 months)
  -This brief cognitive test has participants listen to variable length strings of alphanumeric characters and repeat the characters back verbally in a specific order. They are then scored on the number of correct responses. Scores range from 0 to 21, with higher scores associated with improved cognitive function.
  By doing so, a direct measure of working memory is obtained. Scores on formal testing will be then be analyzed in conjunction with quantification of imaging features (as parceled using DBSI) observed between participants who develop ICANS compared to participants who do not develop ICANs
Changes in cognitive assessment as measured by Hopkins Verbal Learning Test-Received (HVLT-R3) | Baseline, 30 days, 90 days, and 180 days post-transfusion (estimated to be 7 months)
  -This approximately 30 minute long cognitive test has participants learn and free-recall a collection of words from different categories. By doing so, a direct measure of recall and memory is obtained. Scores range from 0 to 30, with higher scores indicating improved cognitive function. Scores on formal testing will be then be analyzed in conjunction with quantification of imaging features (as parceled using DBSI) observed between participants who develop ICANS compared to participants who do not develop ICANs
Changes in cognitive assessment as measured by Montreal-Cognitive Assessment (MocA) | Baseline, 30 days, 90 days, and 180 days post-transfusion (estimated to be 7 months)
  -This approximately 15 minute long cognitive test consists of both written and verbal sections. Participants are scored on the number of correct answers out of 30 (i.e. scores range from 0-30), with higher scores reflecting improved cognitive performance. By doing so, an indirect measure surveying multiple cognitive domains is obtained. Scores on formal testing will be then be analyzed in conjunction with quantification of imaging features (as parceled using DBSI) observed between participants who develop ICANS compared to participants who do not develop ICANs

CONTACTS AND LOCATIONS:
Overall Officials: Armin Ghobadi, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data collected during the trial will be available, after deidentification. This will include the study protocol, statistical analysis plan, and analytic code, beginning 3 months after the start of the study with no end date. This will be made available to researchers who provide a methodologically sound proposal which has been approved by an independent review committee. Interested parties may reach out to Armin Ghobadi, M.D. arminghobadi@wustl.edu
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Beginning 3 months after the start of the study with no end date.
Access Criteria: This will be made available to researchers who provide a methodologically sound proposal which has been approved by an independent review committee. Interested parties may reach out to Armin Ghobadi, M.D. arminghobadi@wustl.edu

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu